CLINICAL TRIAL: NCT02126943
Title: US-based, Observational, Drug Registry of Opsumit® (Macitentan) New Users in Clinical Practice
Brief Title: OPsumit USers Registry
Acronym: OPUS
Status: Completed | Type: Observational
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Other Study IDs: AC-055-503
Record Dates: First submitted 2014-04-29; First posted 2014-04-30 (Estimated); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: PAH; pulmonary arterial hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — macitentan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Opsumit (macitentan): 10 mg tablets
  Interventions: Drug: Opsumit (macitentan)

INTERVENTIONS:
Drug: Opsumit (macitentan) — 10 mg tablets
  Other Names: ACT-064992

SUMMARY:
Prospective observational drug registry developed to characterize the safety profile (including primarily potential serious hepatic risks) and to describe clinical characteristics and outcomes of patients newly treated with Opsumit in the post-marketing setting.

ELIGIBILITY:
Inclusion Criteria:

Patients newly treated with Opsumit defined as a new user of therapy, initiated ≤ 30 days prior to enrollment visit.

Signed ICF

Exclusion Criteria:

Previous user of Opsumit defined as patient who initiated therapy >30 days prior to enrollment.

Patients enrolled in any ongoing clinical trials

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients newly treated with Opsumit
Sampling Method: Non-Probability Sample
Enrollment: 2686 (Actual)
Dates: Start 2014-04-30 (Actual); Primary Completion 2020-04-24 (Actual); Study Completion 2020-04-24 (Actual)

PRIMARY OUTCOMES:
To estimate incidence rates for specified outcomes. | 1 year
  Liver test abnormalities/ Occurrence of Hepatic Adverse Events (HAEs)/ Occurrence of any other AEs/ Discontinuation of Opsumit and reason for stopping therapy/ Hospitalization and death.

SECONDARY OUTCOMES:
To describe demographic and clinical characteristics of patients treated with Opsumit at enrollment and during observation period. | 1 year

OTHER OUTCOMES:
To describe PAH treatment patterns at enrollment and during observation period. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: V McLaughlin, MD, Study Chair — Chair of the OPUS scientific committee (OSC)
Locations (122):
- United States (120):
  - Investigator Site, Mobile, Alabama
  - Investigator Site, Phoenix, Arizona
  - Investigator Site, Fullerton, California
  - Investigator Site, La Jolla, California
  - Investigator Site, Loma Linda, California
  - Investigator Site, Los Angeles, California
  - Investigator Site, Moreno Valley, California
  - Investigator Site, San Juan Capistrano, California
  - Investigator Site, Santa Barbara, California
  - Investigator Site, Stanford, California
  - Investigator Site, Aurora, Colorado
  - Investigator Site, Denver, Colorado
  - Investigator Site, Greeley, Colorado
  - Investigator Site, Wheat Ridge, Colorado
  - Investigator Site, New Haven, Connecticut
  - Investigator Site, Newark, Delaware
  - Investigator Site, Washington D.C., District of Columbia
  - Investigator Site, Brandon, Florida
  - Investigator Site, Celebration, Florida
  - Investigator Site, Clermont, Florida
  - Investigator Site, Fort Lauderdale, Florida
  - Investigator Site, Gainesville, Florida
  - Investigator Site, Hudson, Florida
  - Investigator Site, Jacksonville, Florida
  - Investigator Site, Kissimmee, Florida
  - Investigator Site, Leesburg, Florida
  - Investigator Site, Melbourne, Florida
  - Investigator Site, Miami, Florida
  - Investigator Site, Miami Beach, Florida
  - Investigator Site, Orlando, Florida
  - Investigator Site, Pensacola, Florida
  - Investigator Site, Sebring, Florida
  - Investigator Site, South Miami, Florida
  - Investigator Site, St. Petersburg, Florida
  - Investigator Site, Tampa, Florida
  - Investigator Site, Weston, Florida
  - Investigator Site, Zephyrhills, Florida
  - Investigator Site, Marietta, Georgia
  - Investigator Site, Honolulu, Hawaii
  - Investigator Site, Chicago, Illinois
  - Investigator Site, Oak Brook, Illinois
  - Investigator Site, Carmel, Indiana
  - Investigator Site, Fort Wayne, Indiana
  - Investigator Site, Greenwood, Indiana
  - Investigator Site, Indianapolis, Indiana
  - Investigator Site, Clive, Iowa
  - Investigator Site, Iowa City, Iowa
  - Investigator Site, Kansas City, Kansas
  - Investigator Site, Lexington, Kentucky
  - Investigator Site, Louisville, Kentucky
  - Investigator Site, New Orleans, Louisiana
  - Investigator Site, Shreveport, Louisiana
  - Investigator Site, South Portland, Maine
  - Investigator Site, Baltimore, Maryland
  - Investigator Site, Boston, Massachusetts
  - Investigator Site, Ann Arbor, Michigan
  - Investigator Site, Detroit, Michigan
  - Investigator Site, Lansing, Michigan
  - Investigator Site, Troy, Michigan
  - Investigator Site, Minneapolis, Minnesota
  - Investigator Site, Rochester, Minnesota
  - Investigator Site, St Louis, Missouri
  - Investigator Site, Lincoln, Nebraska
  - Investigator Site, Omaha, Nebraska
  - Investigator Site, Reno, Nevada
  - Investigator Site, Cherry Hill, New Jersey
  - Investigator Site, Newark, New Jersey
  - Investigator Site, Union, New Jersey
  - Investigator Site, Albuquerque, New Mexico
  - Investigator Site, Albany, New York
  - Investigator Site, Brooklyn, New York
  - Investigator Site, Fayetteville, New York
  - Investigator Site, Hauppauge, New York
  - Investigator Site, Mineola, New York
  - Investigator Site, New Hyde Park, New York
  - Investigator Site, New York, New York
  - Investigator Site, The Bronx, New York
  - Investigator Site, Chapel Hill, North Carolina
  - Investigator Site, Durham, North Carolina
  - Investigator Site, Greensboro, North Carolina
  - Investigator Site, Pinehurst, North Carolina
  - Investigator Site, Canton, Ohio
  - Investigator Site, Cincinnati, Ohio
  - Investigator Site, Columbus, Ohio
  - Investigator Site, Dayton, Ohio
  - Investigator Site, Lima, Ohio
  - Investigator Site, Middleburg Heights, Ohio
  - Investigator Site, Toledo, Ohio
  - Investigator Site, Wooster, Ohio
  - Investigator Site, Oklahoma City, Oklahoma
  - Investigator Site, Portland, Oregon
  - Investigator Site, Abington, Pennsylvania
  - Investigator Site, Doylestown, Pennsylvania
  - Investigator Site, Philadelphia, Pennsylvania
  - Investigator Site, Pittsburgh, Pennsylvania
  - Investigator Site, Wynnewood, Pennsylvania
  - Investigator Site, York, Pennsylvania
  - Investigator Site, Anderson, South Carolina
  - Investigator Site, Charleston, South Carolina
  - Investigator Site, Columbia, South Carolina
  - Investigator Site, Rock Hill, South Carolina
  - Investigator Site, Sioux Falls, South Dakota
  - Investigator Site, Chattanooga, Tennessee
  - Investigator Site, Memphis, Tennessee
  - Investigator Site, Dallas, Texas
  - Investigator Site, Houston, Texas
  - Investigator Site, Plano, Texas
  - Investigator Site, San Antonio, Texas
  - Investigator Site, Sherman, Texas
  - Investigator Site, Temple, Texas
  - Investigator Site, Weslaco, Texas
  - Investigator Site, Charlottesville, Virginia
  - Investigator Site, Falls Church, Virginia
  - Investigator Site, Norfolk, Virginia
  - Investigator Site, Richmond, Virginia
  - Investigator Site, Seattle, Washington
  - Investigator Site, Spokane, Washington
  - Investigator Site, Tacoma, Washington
  - Investigator Site, Madison, Wisconsin
  - Investigator Site, Milwaukee, Wisconsin
- Puerto Rico (2):
  - Investigator Site, Ponce, PR
  - Investigator Site, Guaynabo

REFERENCES:
- [Derived] Melendres-Groves LD, Channick RN, Chin KM, McLaughlin VV, MacDonald G, Martin N, Ong R, Sandros M, Kim NH. Characteristics, Treatment Patterns and Outcomes of Patients with Pulmonary Arterial Hypertension by Race and Ethnicity Using Real-World Data from the Combined OPUS/OrPHeUS Studies. Adv Ther. 2025 Nov 19. doi: 10.1007/s12325-025-03403-4. Online ahead of print. PMID 41258625
- [Derived] Kim NH, Chin KM, McLaughlin VV, Ong R, MacDonald G, Martin N, Senatore A, Channick R. Macitentan and Tadalafil Combination Therapy in Patients with Pulmonary Arterial Hypertension and Cardiovascular Comorbidities: Real-World Evidence from OPUS and OrPHeUS. Adv Ther. 2025 Jul;42(7):3306-3333. doi: 10.1007/s12325-025-03180-0. Epub 2025 May 19. PMID 40388087
- [Derived] Chin KM, Channick R, Kim NH, Ong R, Turricchia S, Martin N, Mitchell L, McLaughlin VV. Macitentan in Pulmonary Arterial Hypertension Due to Congenital Heart Disease (CHD-PAH): Real-World Evidence from the OPUS/OrPHeUS Studies. Cardiol Ther. 2024 Dec;13(4):775-796. doi: 10.1007/s40119-024-00386-1. Epub 2024 Nov 25. PMID 39585521
- [Derived] Channick R, Chin KM, McLaughlin VV, Lammi MR, Zamanian RT, Turricchia S, Ong R, Mitchell L, Kim NH. Macitentan in Pulmonary Arterial Hypertension Associated with Connective Tissue Disease (CTD-PAH): Real-World Evidence from the Combined OPUS/OrPHeUS Dataset. Cardiol Ther. 2024 Jun;13(2):315-339. doi: 10.1007/s40119-024-00361-w. Epub 2024 Mar 7. PMID 38451426
- [Derived] Kim NH, Chin KM, McLaughlin VV, DuBrock H, Restrepo-Jaramillo R, Safdar Z, MacDonald G, Martin N, Rosenberg D, Solonets M, Channick R. Safety of Macitentan for the Treatment of Portopulmonary Hypertension: Real-World Evidence from the Combined OPUS/OrPHeUS Studies. Pulm Ther. 2024 Mar;10(1):85-107. doi: 10.1007/s41030-023-00251-x. Epub 2024 Jan 7. PMID 38184507